CLINICAL TRIAL: NCT05187468
Title: The Effectiveness of Radial Extracorporeal Shockwave on Upper Trapezius Myofascial Trigger Points
Brief Title: The Effectiveness of Radial ESWT on Upper Trapezius Mtrps
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: European University Cyprus (Other)
Responsible Party: Principal Investigator, Rentzias Panagiotis, Lecturer, European University Cyprus
Allocation: Randomized | Model: Sequential | Masking: Triple | Purpose: Treatment
Other Study IDs: EuropeanUC
Record Dates: First submitted 2021-09-19; First posted 2022-01-11 (Actual); Last update posted 2022-01-11 (Actual); Status verified 2021-09

CONDITIONS: Myofascial Pain Syndrome; Myofascial Trigger Point Pain; Upper Trapezius Trigger Points
Keywords: Myofascial Trigger points; upper trapezius; Myofascial pain syndrome; Mtrps
MeSH Terms: conditions — Myofascial Pain Syndromes | interventions — Extracorporeal Shockwave Therapy; Ultrasonic Therapy; Massage

STUDY DESIGN:
Who Masked: Participant, Care Provider, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- ESWT 1 (Experimental): Extracorporeal Shockwave Therapy 1000 pulses, 60 mJ, 10 Hz
  Interventions: Device: Extracorporeal Shockwave Therapy
- ESWT 2 (Experimental): Extracorporeal Shockwave Therapy 2000 pulses, 60 mJ, 10 Hz
  Interventions: Device: Extracorporeal Shockwave Therapy
- Ultrasound therapy, Massage, Heat Pack (Active Comparator): 10 Min massage 5 min US therapy 10 min Heat pack
  Interventions: Device: Ultrasound therapy, Massage, Heat pack

INTERVENTIONS:
Device: Extracorporeal Shockwave Therapy — 1000 pulses at 60 mj, 10 Hz
  Other Names: ESWT; rSWT
  Arms: ESWT 1
Device: Extracorporeal Shockwave Therapy — 2000 pulses at 60 mj, 10 Hz
  Arms: ESWT 2
Device: Ultrasound therapy, Massage, Heat pack — Ultrasound therapy 5 min, 1,2W/cm2, 10 min Massage, 10 min heat pack
  Arms: Ultrasound therapy, Massage, Heat Pack

SUMMARY:
This study looked after the effectiveness of radial ESWT on upper trapezius mtrps. There were three intervention groups which recieved either ESWT or standard care. VAS, PPT, Neck ROM and Cervical functionality were the main outcomes.

DETAILED DESCRIPTION:
This study was a randomized controlled trial consisted of three intervention groups. Two of them recieved ESWT with different parameters in each group, while the third one was standard care recieving Ultrasound therapy, Therapeutic massage and Heat packs Participants were divided randomly into the three groups. Participants were blind to the group allocated and also the therapist and outcome investigator were blind.

The participants recieved three weekly sessions. The evaluation took place before therapy, after each session and one month after last session.

The outcome measures was the pain intensity with VAS, the pain tolerance to pressure by an algometer device, the range of motion of neck measured by electronic goniometer and and functionality of neck measured by the Northwick Park Neck Pain

ELIGIBILITY:
Inclusion Criteria:

* Pain between shoulder and neck on upper trapezius muscle
* Three out of five of Travel and Simons criteria for myofascial trigger points

Exclusion Criteria:

* Fibromyalgia diagnosis
* Systemic diseases diagnosis,
* Pacemaker, under 18,
* Any kind of cervical disorder or surgery,
* Mental disorders

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 56 (Actual)
Dates: Start 2019-08-01 (Actual); Primary Completion 2019-10-30 (Actual); Study Completion 2020-02-28 (Actual)

PRIMARY OUTCOMES:
Pain intensity on myofascial trigger points | baseline
  Visual Analogue Scale 1-10 (1 is the least pain, 10 is the worst pain)
Pain intensity on myofascial trigger points | one week
  Visual Analogue Scale 1-10 (1 is the least pain, 10 is the worst pain)
Pain intensity on myofascial trigger points | two weeks
  Visual Analogue Scale 1-10 (1 is the least pain, 10 is the worst pain)
Pain intensity on myofascial trigger points | three weeks
  Visual Analogue Scale 1-10 (1 is the least pain, 10 is the worst pain)
Pain intensity on myofascial trigger points | 1 month after
  Visual Analogue Scale 1-10 (1 is the least pain, 10 is the worst pain)
Pressure Pain Threshold | baseline
  Pain tolerance to compression. Measured in kilos
Pressure Pain Threshold | one week
  Pain tolerance to compression. Measured in kilos
Pressure Pain Threshold | two weeks
  Pain tolerance to compression. Measured in kilos
Pressure Pain Threshold | three weeks
  Pain tolerance to compression. Measured in kilos
Pressure Pain Threshold | one month after
  Pain tolerance to compression. Measured in kilos
cervical range of motion | baseline
  Goniometer (measured in degrees)
cervical range of motion | one week
  Goniometer (measured in degrees)
cervical range of motion | two weeks
  Goniometer (measured in degrees)
cervical range of motion | three weeks
  Goniometer (measured in degrees)
cervical range of motion | one month after
  Goniometer (measured in degrees)
Northwick Park Neck Pain questionnaire | baseline
  functionality of Neck related to pain for daily activities. measured in % (36 questions). Higher the %, greater the disability
Northwick Park Neck Pain questionnaire | one week
  functionality of Neck related to pain for daily activities. measured in % (36 questions). Higher the %, greater the disability
Northwick Park Neck Pain questionnaire | two weeks
  functionality of Neck related to pain for daily activities. measured in % (36 questions). Higher the %, greater the disability
Northwick Park Neck Pain questionnaire | three weeks
  functionality of Neck related to pain for daily activities. measured in % (36 questions). Higher the %, greater the disability
Northwick Park Neck Pain questionnaire | one month after
  functionality of Neck related to pain for daily activities. measured in % (36 questions). Higher the %, greater the disability

CONTACTS AND LOCATIONS:
Locations (1):
- European University Cyprus, Nicosia, Cyprus